CLINICAL TRIAL: NCT01336725
Title: Learning and Coping With Chronic Illness
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: May Solveig Fagermoen/Nurse researcher, Oslo university hospital
Other Study IDs: S-08662c 2008/17575 (REK)
Record Dates: First submitted 2011-04-14; First posted 2011-04-18 (Estimated); Last update posted 2011-04-18 (Estimated); Status verified 2011-04

CONDITIONS: Morbid Obesity
Keywords: Morbid obesity; Patient education
MeSH Terms: conditions — Obesity, Morbid | interventions — Educational Status

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Morbid obesity: All attending learning and mastery courses for persons with morbid obesity
  Interventions: Behavioral: Teaching life style changes; Other: Active participation; Other: Teaching

INTERVENTIONS:
Behavioral: Teaching life style changes — Single group: Teaching, group sessions, physical activity
Other: Active participation — Obesity group attend 10 group sessions,are informed about and discuss needed life style changes such as weight loss and participate in physical activity and cooking.
Other: Teaching — Morbid obesity group attend 40 hours of group sessions

SUMMARY:
The purpose of this study is to determine whether the participants have improved their scores on health related quality of life (HRQL) 1 year after completing a learning and mastery course and whether sociodemographic variables are associated with HRQL.

DETAILED DESCRIPTION:
Persons with chronic illnesses have to adjust to changes in their life-style. In the last 10 years Learning and Mastery Centres have been established in Norwegian hospitals to offer patient education for the chronically ill. It is not known whether these courses impact any changes in HRQL 1 year after course completion.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of morbid obesity
* attending learning and mastery course for the obese

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Learning and mastery centre
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2009-01; Primary Completion 2010-09 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Health related quality of life | 1 year after course completion

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo universiy hospital, Aker, Oslo, Norway

REFERENCES:
- [Derived] Lerdal A, Gay CL, Bonsaksen T, Fagermoen MS. Predictors of physical and mental health in persons with morbid obesity attending a patient education course - a two-year follow-up study. Health Qual Life Outcomes. 2017 May 15;15(1):103. doi: 10.1186/s12955-017-0675-z. PMID 28506306
- [Derived] Andenaes R, Fagermoen MS, Eide H, Lerdal A. Changes in health-related quality of life in people with morbid obesity attending a learning and mastery course. A longitudinal study with 12-months follow-up. Health Qual Life Outcomes. 2012 Aug 18;10:95. doi: 10.1186/1477-7525-10-95. PMID 22901031